CLINICAL TRIAL: NCT03949296
Title: A Randomized, Placebo-Controlled Study of Mindfulness Meditation in Treating Insomnia in Multiple Sclerosis
Brief Title: Mindfulness Meditation in Treating Insomnia in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Griffin Hospital (Other)
Collaborators: Yale-Griffin Prevention Research Center (Other); Yale University- Stress Center (Unknown)
Responsible Party: Principal Investigator, Joseph B. Guarnaccia, Director of the MS Treatment Center at Griffin Hospital, Griffin Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2017-01
Record Dates: First submitted 2018-12-29; First posted 2019-05-14 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Insomnia Chronic; Multiple Sclerosis
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: A placebo-controlled, randomized, single-blinded clinical study involving a projected 90 participants with multiple sclerosis in a 50:50 randomization scheme.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Intervention (Active Comparator): Mindfulness-Based Treatment for Insomnia intervention led by a certified instructor. It is adapted from the Mindfulness-Based Stress Reduction Curriculum developed by the Center for Mindfulness in Medicine, Health Care, and Society at the University of Massachusetts Medical School. It introduces the concept of mindfulness and provides the opportunity to practice it within sessions and during home practice. Participants learn about stress, and explore habitual behavioral, physical, emotional and cognitive patterns, as well as more effective responses to challenges and demands of everyday life. Each class includes mindfulness practice, group discussions, and practices and exercises related to the class topics. Participants receive home assignments with guided meditation and yoga practices.
  Interventions: Behavioral: Mindfulness Intervention
- Sleep Hygiene (Placebo Comparator): Control group participants attend a 30-minute group counseling session on sleep hygiene. The session includes a handout from the Centre for Clinical Intervention in Australia that provides 15 sleep hygiene tips.
  Interventions: Behavioral: Sleep Hygiene

INTERVENTIONS:
Behavioral: Mindfulness Intervention — 10-session program
  1. Introduction to mindfulness and its potential benefits
  2. Introduction to mindful practices and yoga poses
  3. Conditioned reactions to stress; integrating mindfulness into everyday life
  4. Challenges and insights gained in practicing mindfulness
  5. Using mindfulness to observe and reduce negative means of reacting to stress, and find more effective responses
  6. Reacting vs. responding to stressors
  7. Self-regulation and coping with stressors and communication challenges
  8. Fostering continuity of moment-to-moment awareness while practicing different forms of mindfulness
  9. Choosing and creating one's own blend of mindfulness practices
  10. Maintaining momentum to practice mindfulness once the program ends
  Arms: Mindfulness Intervention
Behavioral: Sleep Hygiene — Session includes a handout with15 sleep hygiene tips:
  1. Maintain a regular sleep pattern
  2. Only try to sleep when feeling tired or sleepy
  3. If unable to sleep, do something calm until feeling tired and returning to bed
  4. Avoid caffeine & nicotine for 4-6 hours before going to bed
  5. Avoid alcohol for 4-6 hours before going to bed
  6. Use the bed only for sleeping and sex
  7. Avoid naps during the day
  8. Develop rituals to get relaxed and ready to sleep
  9. Try a hot bath prior to bedtime
  10. Avoid checking the clock during the night
  11. Use a sleep diary for a few weeks to track progress
  12. Avoid strenuous exercise before bedtime
  13. Avoid a heavy meal before bedtime
  14. Create a sleep environment that is quiet, comfortable, and dark
  15. Maintain a regular daytime routine
  Arms: Sleep Hygiene

SUMMARY:
Purpose To determine whether Mindfulness-Based Treatment for Insomnia (MBTI) is more effective in the treatment of chronic insomnia disorder (CID) in patients with multiple sclerosis (MS) when compared with standard sleep hygiene counseling.

Specific Aims / Hypotheses

Our specific aims are to determine:

* Whether MBTI is more effective than standard sleep hygiene counseling in improving objectively-measured sleep quality among this group of MS patients with CID, as measured by the Fitbit Charge 2 activity tracker.
* Whether MBTI is more effective than standard sleep hygiene counseling in improving self-reported sleep quality among this group of MS patients with CID, as measured by the Pittsburgh Sleep Quality Index (PSQI).
* Whether MTBI is more effective than standard sleep hygiene counseling in reducing self-reported severity of insomnia among this group of MS patients with CID, as measured by the Insomnia Severity Index (ISI).
* Whether MBTI is more effective than standard sleep hygiene counseling in improving self-reported quality of life among this group of MS patients with CID, as measured by the Multiple Sclerosis Quality of Life Inventory (MSQLI).

We hypothesize that among study participants with MS and CID:

* MBTI will improve their objectively-measured sleep quality, as measured by the Fitbit Charge 2 activity tracker.
* MBTI will improve their self-reported sleep quality, as measured by the PSQI.
* MBTI will reduce their self-reported severity of insomnia, as measured by the ISI.
* Improvement in sleep quality and reduction in insomnia severity will result in improvement in self-reported quality of life, as measured by MSQLI scores.
* MBTI will be superior to sleep hygiene counseling in improving sleep quality, reducing insomnia severity, and improving quality of life.

DETAILED DESCRIPTION:
BACKGROUND:

An estimated 25 to 40 percent of individuals with multiple sclerosis (MS) suffer from chronic insomnia, and the prevalence of sleep disorders is often unrecognized. Chronic insomnia disorder (CID) is defined as persistent difficulty with sleep initiation, duration, consolidation, or quality that occurs despite adequate opportunity and circumstances for sleep, leading to daytime impairment, and ongoing for at least three consecutive months.

Common causes of CID in MS include motor disorders such as cramps, spasms, restless leg syndrome and periodic limb movements, neuropathic pain, bladder dysfunction (such as nocturia), and obstructive sleep apnea. Depression, anxiety, daytime fatigue, and cognitive dysfunction are also associated with sleep disorders in MS. Moreover, treatments for the underlying disease, such as interferon therapy, as well as treatments for various symptoms of MS, such as stimulant medications used to treat fatigue, may also contribute to insomnia.

Many patients manage their insomnia using benzodiazepines and other medications, which may be associated with a number of adverse effects, including dependence and tolerance, cognitive dysfunction, and depression. Furthermore, other adverse effects of benzodiazepines arise from their use in combination with other drugs such as opioid narcotics for pain. Therefore, it is desirable to find effective nonpharmacological treatments for insomnia in patients with multiple sclerosis.

Psychologically-based and behavioral treatments have been widely tested in various cohorts of patients with CID with and without co-morbid conditions. These methods include cognitive behavioral therapies (CBT), sleep hygiene programs, mindfulness meditation, and others. In a randomized controlled clinical trial of 72 women with CID and MS in Iran, CBT treatment was associated with improved sleep quality as measured by the Pittsburgh Sleep Quality Index (PSQI). A case series of 11 patients with chronic insomnia and MS who were treated with CBT at the Cleveland Clinic Sleep Disorders Center improved on measures of insomnia, fatigue and depression, as well as an increase in total sleep time of 1.5 hours.

Mindfulness based stress reduction (MBSR) is an empirically-supported intervention designed to decrease stress, chronic and acute pain and anxiety in adults. Mindfulness is the practice of focusing full attention on the present moment intentionally and without judgment. The practice of mindfulness is hypothesized to reduce feelings of distress and stress reactivity by increasing one's awareness of and ability to tolerate thoughts and emotions. Mindfulness may help individuals decrease distress and over-reactivity to events and increase the ability to respond to events in ways that one consciously chooses (rather than through automatic 'mindless" behaviors). Mindfulness-based interventions such as MBSR teach mindfulness through meditation, yoga, present-minded awareness in everyday life, and discussions of stress physiology and coping.

Several studies have demonstrated the effectiveness of MBSR interventions in the treatment of insomnia. Long-term meditators have been shown to have increased parietal-occipital gamma (25-40 Hz) during NREM (non-rapid eye movement sleep), showing that MBSR can induce objective changes in sleep architecture. MBSR and MBTI (mindfulness based treatment of insomnia) have been shown in randomized, controlled studies to decrease sleep latency and total waking time and increase sleep time.These effects, moreover, have been durable. However, a meta-analysis of 6 randomized controlled trials involving 330 participants showed that mindfulness meditation significantly improved total wake time and sleep quality, but had no significant effects on sleep onset latency, total sleep time, wake after sleep onset, sleep efficiency, total wake time, Insomnia Severity Index (ISI), PSQI, or Dysfunctional Beliefs and Attitudes Sleep Scale (DBAS).

Mindfulness training has been shown to be beneficial in improving several symptoms of MS, including those that have been shown to impact sleep. A randomized, controlled study of 150 patients undergoing mindfulness training showed improvements in quality of life and well-being, including fatigue and depression. Furthermore, there is Class 1 evidence that stress reduction in MS can affect the underlying inflammatory biology of MS, as evidenced by a reduction in new MRI lesions. However, many other studies showing benefits of stress reduction in MS are limited by their descriptive nature and non-controlled design.

The significance of this study is that while there are data showing the effectiveness of mindfulness-based techniques in treating insomnia in general, and some data showing the benefits of using non-mindfulness stress reduction techniques in the management of MS-related insomnia, there have been no studies to date on the efficacy of mindfulness techniques in treating MS-related insomnia.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women age 18 years or older
2. Diagnosis of multiple sclerosis per the 2014 Revised MacDonald criteria
3. Moderate to severe insomnia based on Insomnia Severity Index score
4. Kurtzke Expanded Disability Status Scale (EDSS) score between 0 and 7.0
5. Stable medications and disease activity for the past 30 days
6. Willingness to visit Griffin Hospital for up to 13 times if assigned to the mindfulness group, or up to 4 times if assigned to the sleep hygiene group, for study assessment and counseling or educational sessions

Exclusion Criteria:

1. Diagnosis of obstructive sleep apnea or narcolepsy
2. High risk of obstructive sleep apnea, as determined by the STOP-Bang questionnaire, if no known diagnosis of sleep apnea
3. Significant pulmonary, cardiac, hepatic or other medical conditions
4. Relapse of MS symptoms within the 30 days prior to study entry
5. Use of corticosteroids, either IV or oral, for exacerbations of symptoms
6. Inability to comply with the protocol
7. A lack of proficiency in reading, writing in, and understanding English
8. Body mass index (BMI) > 39 (350 lb. due to the limitations of the scale used for the study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
Sleep Quality | 4 months
  Objective sleep quality will be measured using a Fitbit Charge activity monitor to be worn daily during the 10-week intervention, and daily during a 4-month post-intervention period. For the purpose of assessing the impact of the intervention on objective sleep quality, the first week of Fitbit sleep data collected during the 10-week intervention (i.e., during the week of the mindfulness orientation session) will count as baseline data; the last week of the 10-week intervention will count as post-intervention data; and the last week of the 4-month post-intervention period will be used to assess the sustainability of the intervention. Data from the remaining weeks of the 10-week intervention and 4-month post-intervention periods will be used to examine whether participants experience an upward trend in sleep quality during the course of the study.

SECONDARY OUTCOMES:
Self-Reported Sleep Quality | 4 months
  Self-reported sleep quality will be measured using the Pittsburgh Sleep Quality Index (PSQI) at baseline, at the end of the 10-week intervention, and at 4 months post-intervention. The PSQI is a self-rated questionnaire to assess perceived sleep quality and disturbances over a 1-month time interval. This 19-item instrument uses a Likert scale (ranging from 0 to 3) to assess 7 clinically derived domains of sleep: sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these 7 components yields one global score. Clinical and clinimetric properties of the PSQI were assessed over an 18-month period with "good" vs. "poor" sleepers. A global score > 5 yielded a diagnostic sensitivity of 89.6% and specificity of 86.5% (kappa = 0.75, p < 0.001) in distinguishing good vs. poor sleepers.
Self-Reported Quality of Life | 4 months
  Self-reported quality of life will be measured at baseline, the end of the 10-week intervention, and 4 months post-intervention using the Multiple Sclerosis Quality of Life Index (MSQLI). The MSQLI includes a set of 10 questionnaires to provide a quality of life measure that is both generic and MS-specific. The questionnaires assess health status, fatigue, pain, sexual satisfaction, bladder control, bowel control, visual impairment, perceived deficits, mental health, and social support. Each individual scale generates a separate score. There is no global composite combining all the scales into a single score. There is good internal consistency reliability for the subscales of the MSQLI, with the lowest alpha being 0.67 (for social functioning on SF-36). Other coefficients range from 0.78 (BWCS) to 0.97 (MSSS). Test-retest reliability on the SF-36 ranges from 0.60 (social functioning) to 0.81 (physical functioning).

OTHER OUTCOMES:
Adverse Events | 4 months
  Any adverse events, including relapse of MS, experienced by study participants will be noted at the end of the 10-week intervention, and at 4-months post-intervention. In addition, if participants report any adverse events by contacting the research staff and/or study PI at any other time points during the study, these will be noted as well. The study team will address the handling of adverse events on a case-by-case basis.
Progression of MS | 4 months
  Progression of MS will be measured by administering the Kurtzke Expanded Disability Status Scale (EDSS) at baseline (clinical screening), the end of the 10-week intervention, and 4 months post-intervention. The EDSS is a method of quantifying the degree of neurologic impairment in MS patients. It quantifies disability in 8 Functional Systems (pyramidal, cerebellar, brainstem, sensory, bowel and bladder, visual, cerebral, and "other"), and allows neurologists or other trained examiners to assign a Functional System Score (FSS) in each FS. Each FSS is an ordinal clinical rating scale ranging from 0 to 5 or 6. The EDSS is an ordinal clinical rating scale ranging from 0 (normal neurologic examination) to 10 (death due to MS) in half-point increments.
Muscle Spasticity | 4 months
  Since muscle spasticity is a frequent cause of insomnia in MS patients, the Modified Ashworth Scale (MAS) will be used to characterize the degree of spasticity at baseline (clinical screening), the end of the 10-week intervention and 4 months post-intervention among members of our study population. The MAS is a clinician-administered measure of muscle spasticity in patients with MS or other conditions such as stroke or spinal cord injury. It involves a subjective clinical assessment, without the use of specialized equipment, of muscle resistance to passive range of motion (ROM) about a single joint, while a patient is in a supine position. It uses a nominal scale ranging from 0 (no resistance) to 4 (rigidity), with a 1+ scoring category added to indicate resistance through less than half of the movement.
Restless Leg | 4 months
  Since restless leg syndrome can impact insomnia in MS patients, self-reported restless legs syndrome severity will be measured using the International Restless Legs Scale (IRLS) at baseline, at the end of the 10-week intervention, and 4 months post-intervention to characterize the extent of this condition in our study population. The IRLS was developed by the International RLS Study Group to measure perceived severity of restless legs syndrome in the past week prior to administration. It includes 10 questions addressing respondents' perceptions of RLS-related discomfort, need to move around, relief from moving around, severity of sleep disturbance and tiredness from RLS symptoms, severity of RLS as a whole, frequency and severity of symptoms, severity of impact on daily living, and severity of mood disturbance. Response options are based on a 5-point scale ranging from 0 to 4, with 4 being very severe.
Medication and Supplements | 4 months
  A list of medications and/or supplements used will be collected at baseline, the end of the 10-week intervention, and 4-months post-intervention to track changes in use of medication or supplements during the course of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph B Guarnaccia, MD, Principal Investigator — Griffin Hospital
Locations (1):
- Yale-Griffin Prevention Research Center, Derby, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Viana P, Rodrigues E, Fernandes C, Matas A, Barreto R, Mendonca M, Peralta R, Geraldes R. InMS: Chronic insomnia disorder in multiple sclerosis - a Portuguese multicentre study on prevalence, subtypes, associated factors and impact on quality of life. Mult Scler Relat Disord. 2015 Sep;4(5):477-483. doi: 10.1016/j.msard.2015.07.010. Epub 2015 Jul 26. PMID 26346798
- [Background] Veauthier C, Radbruch H, Gaede G, Pfueller CF, Dorr J, Bellmann-Strobl J, Wernecke KD, Zipp F, Paul F, Sieb JP. Fatigue in multiple sclerosis is closely related to sleep disorders: a polysomnographic cross-sectional study. Mult Scler. 2011 May;17(5):613-22. doi: 10.1177/1352458510393772. Epub 2011 Jan 28. PMID 21278050
- [Background] Veauthier C, Paul F. Sleep disorders in multiple sclerosis and their relationship to fatigue. Sleep Med. 2014 Jan;15(1):5-14. doi: 10.1016/j.sleep.2013.08.791. Epub 2013 Nov 15. PMID 24360534
- [Background] Braley TJ, Segal BM, Chervin RD. Obstructive sleep apnea and fatigue in patients with multiple sclerosis. J Clin Sleep Med. 2014 Feb 15;10(2):155-62. doi: 10.5664/jcsm.3442. PMID 24532998
- [Background] Brass SD, Li CS, Auerbach S. The underdiagnosis of sleep disorders in patients with multiple sclerosis. J Clin Sleep Med. 2014 Sep 15;10(9):1025-31. doi: 10.5664/jcsm.4044. PMID 25142763
- [Background] Cartwright RD. Alcohol and NREM parasomnias: evidence versus opinions in the international classification of sleep disorders, 3rd edition. J Clin Sleep Med. 2014 Sep 15;10(9):1039-40. doi: 10.5664/jcsm.4050. No abstract available. PMID 25221449
- [Background] Merlino G, Fratticci L, Lenchig C, Valente M, Cargnelutti D, Picello M, Serafini A, Dolso P, Gigli GL. Prevalence of 'poor sleep' among patients with multiple sclerosis: an independent predictor of mental and physical status. Sleep Med. 2009 Jan;10(1):26-34. doi: 10.1016/j.sleep.2007.11.004. Epub 2008 Jan 22. PMID 18207453
- [Background] Stanton BR, Barnes F, Silber E. Sleep and fatigue in multiple sclerosis. Mult Scler. 2006 Aug;12(4):481-6. doi: 10.1191/135248506ms1320oa. PMID 16900762
- [Background] Boe Lunde HM, Aae TF, Indrevag W, Aarseth J, Bjorvatn B, Myhr KM, Bo L. Poor sleep in patients with multiple sclerosis. PLoS One. 2012;7(11):e49996. doi: 10.1371/journal.pone.0049996. Epub 2012 Nov 14. PMID 23166808
- [Background] Bamer AM, Johnson KL, Amtmann DA, Kraft GH. Beyond fatigue: Assessing variables associated with sleep problems and use of sleep medications in multiple sclerosis. Clin Epidemiol. 2010 May 1;2010(2):99-106. doi: 10.2147/CLEP.S10425. PMID 20838467
- [Background] Italian REMS Study Group; Manconi M, Ferini-Strambi L, Filippi M, Bonanni E, Iudice A, Murri L, Gigli GL, Fratticci L, Merlino G, Terzano G, Granella F, Parrino L, Silvestri R, Arico I, Dattola V, Russo G, Luongo C, Cicolin A, Tribolo A, Cavalla P, Savarese M, Trojano M, Ottaviano S, Cirignotta F, Simioni V, Salvi F, Mondino F, Perla F, Chinaglia G, Zuliani C, Cesnik E, Granieri E, Placidi F, Palmieri MG, Manni R, Terzaghi M, Bergamaschi R, Rocchi R, Ulivelli M, Bartalini S, Ferri R, Lo Fermo S, Ubiali E, Viscardi M, Rottoli M, Nobili L, Protti A, Ferrillo F, Allena M, Mancardi G, Guarnieri B, Londrillo F. Multicenter case-control study on restless legs syndrome in multiple sclerosis: the REMS study. Sleep. 2008 Jul;31(7):944-52. PMID 18655317
- [Background] Braley TJ, Segal BM, Chervin RD. Sleep-disordered breathing in multiple sclerosis. Neurology. 2012 Aug 28;79(9):929-36. doi: 10.1212/WNL.0b013e318266fa9d. Epub 2012 Aug 15. PMID 22895593
- [Background] Pokryszko-Dragan A, Bilinska M, Gruszka E, Biel L, Kaminska K, Konieczna K. Sleep disturbances in patients with multiple sclerosis. Neurol Sci. 2013 Aug;34(8):1291-6. doi: 10.1007/s10072-012-1229-0. Epub 2012 Oct 30. PMID 23109097
- [Background] Mendozzi L, Tronci F, Garegnani M, Pugnetti L. Sleep disturbance and fatigue in mild relapsing remitting multiple sclerosis patients on chronic immunomodulant therapy: an actigraphic study. Mult Scler. 2010 Feb;16(2):238-47. doi: 10.1177/1352458509354551. Epub 2009 Dec 22. PMID 20028705
- [Background] Lanza G, Ferri R, Bella R, Ferini-Strambi L. The impact of drugs for multiple sclerosis on sleep. Mult Scler. 2017 Jan;23(1):5-13. doi: 10.1177/1352458516664034. Epub 2016 Aug 19. PMID 27503906
- [Background] Siebern AT, Manber R. Insomnia and its effective non-pharmacologic treatment. Med Clin North Am. 2010 May;94(3):581-91. doi: 10.1016/j.mcna.2010.02.005. PMID 20451034
- [Background] Martires J, Zeidler M. The value of mindfulness meditation in the treatment of insomnia. Curr Opin Pulm Med. 2015 Nov;21(6):547-52. doi: 10.1097/MCP.0000000000000207. PMID 26390335
- [Background] Gong H, Ni CX, Liu YZ, Zhang Y, Su WJ, Lian YJ, Peng W, Jiang CL. Mindfulness meditation for insomnia: A meta-analysis of randomized controlled trials. J Psychosom Res. 2016 Oct;89:1-6. doi: 10.1016/j.jpsychores.2016.07.016. Epub 2016 Jul 26. PMID 27663102
- [Background] Abbasi S Ms, Alimohammadi N PhD, Pahlavanzadeh S Ms. Effectiveness of Cognitive Behavioral Therapy on the Quality of Sleep in Women with Multiple Sclerosis: A Randomized Controlled Trial Study. Int J Community Based Nurs Midwifery. 2016 Oct;4(4):320-328. PMID 27713895
- [Background] Clancy M, Drerup M, Sullivan AB. Outcomes of Cognitive-Behavioral Treatment for Insomnia on Insomnia, Depression, and Fatigue for Individuals with Multiple Sclerosis: A Case Series. Int J MS Care. 2015 Nov-Dec;17(6):261-7. doi: 10.7224/1537-2073.2014-071. PMID 26664331
- [Background] Kabat-Zinn J (1990). Full Catastrophe Living. New York. NY. Bantam Books
- [Background] Ferrarelli F, Smith R, Dentico D, Riedner BA, Zennig C, Benca RM, Lutz A, Davidson RJ, Tononi G. Experienced mindfulness meditators exhibit higher parietal-occipital EEG gamma activity during NREM sleep. PLoS One. 2013 Aug 28;8(8):e73417. doi: 10.1371/journal.pone.0073417. eCollection 2013. PMID 24015304
- [Background] Britton WB, Haynes PL, Fridel KW, Bootzin RR. Mindfulness-based cognitive therapy improves polysomnographic and subjective sleep profiles in antidepressant users with sleep complaints. Psychother Psychosom. 2012;81(5):296-304. doi: 10.1159/000332755. Epub 2012 Jul 20. PMID 22832540
- [Background] Britton WB, Haynes PL, Fridel KW, Bootzin RR. Polysomnographic and subjective profiles of sleep continuity before and after mindfulness-based cognitive therapy in partially remitted depression. Psychosom Med. 2010 Jul;72(6):539-48. doi: 10.1097/PSY.0b013e3181dc1bad. Epub 2010 May 13. PMID 20467003
- [Background] Grossman P, Kappos L, Gensicke H, D'Souza M, Mohr DC, Penner IK, Steiner C. MS quality of life, depression, and fatigue improve after mindfulness training: a randomized trial. Neurology. 2010 Sep 28;75(13):1141-9. doi: 10.1212/WNL.0b013e3181f4d80d. PMID 20876468
- [Background] Simpson R, Booth J, Lawrence M, Byrne S, Mair F, Mercer S. Mindfulness based interventions in multiple sclerosis--a systematic review. BMC Neurol. 2014 Jan 17;14:15. doi: 10.1186/1471-2377-14-15. PMID 24438384
- [Background] Mohr DC, Lovera J, Brown T, Cohen B, Neylan T, Henry R, Siddique J, Jin L, Daikh D, Pelletier D. A randomized trial of stress management for the prevention of new brain lesions in MS. Neurology. 2012 Jul 31;79(5):412-9. doi: 10.1212/WNL.0b013e3182616ff9. Epub 2012 Jul 11. PMID 22786596
- [Background] Reynard AK, Sullivan AB, Rae-Grant A. A systematic review of stress-management interventions for multiple sclerosis patients. Int J MS Care. 2014 Fall;16(3):140-4. doi: 10.7224/1537-2073.2013-034. PMID 25337056
- [Background] Dias RA, Hardin KA, Rose H, Agius MA, Apperson ML, Brass SD. Sleepiness, fatigue, and risk of obstructive sleep apnea using the STOP-BANG questionnaire in multiple sclerosis: a pilot study. Sleep Breath. 2012 Dec;16(4):1255-65. doi: 10.1007/s11325-011-0642-6. Epub 2012 Jan 21. PMID 22270686
- [Background] Tan A, Yin JD, Tan LW, van Dam RM, Cheung YY, Lee CH. Predicting obstructive sleep apnea using the STOP-Bang questionnaire in the general population. Sleep Med. 2016 Nov-Dec;27-28:66-71. doi: 10.1016/j.sleep.2016.06.034. Epub 2016 Oct 27. PMID 27938922
- [Background] Chiu HY, Chen PY, Chuang LP, Chen NH, Tu YK, Hsieh YJ, Wang YC, Guilleminault C. Diagnostic accuracy of the Berlin questionnaire, STOP-BANG, STOP, and Epworth sleepiness scale in detecting obstructive sleep apnea: A bivariate meta-analysis. Sleep Med Rev. 2017 Dec;36:57-70. doi: 10.1016/j.smrv.2016.10.004. Epub 2016 Nov 5. PMID 27919588
- [Background] Abrishami A, Khajehdehi A, Chung F. A systematic review of screening questionnaires for obstructive sleep apnea. Can J Anaesth. 2010 May;57(5):423-38. doi: 10.1007/s12630-010-9280-x. Epub 2010 Feb 9. PMID 20143278
- [Background] https://www.fitbit.com/charge2
- [Background] Ancoli-Israel S, Cole R, Alessi C, Chambers M, Moorcroft W, Pollak CP. The role of actigraphy in the study of sleep and circadian rhythms. Sleep. 2003 May 1;26(3):342-92. doi: 10.1093/sleep/26.3.342. PMID 12749557
- [Background] Van de Water AT, Holmes A, Hurley DA. Objective measurements of sleep for non-laboratory settings as alternatives to polysomnography--a systematic review. J Sleep Res. 2011 Mar;20(1 Pt 2):183-200. doi: 10.1111/j.1365-2869.2009.00814.x. PMID 20374444
- [Background] de Zambotti M, Baker FC, Willoughby AR, Godino JG, Wing D, Patrick K, Colrain IM. Measures of sleep and cardiac functioning during sleep using a multi-sensory commercially-available wristband in adolescents. Physiol Behav. 2016 May 1;158:143-9. doi: 10.1016/j.physbeh.2016.03.006. Epub 2016 Mar 9. PMID 26969518
- [Background] Lee HA, Lee HJ, Moon JH, Lee T, Kim MG, In H, Cho CH, Kim L. Comparison of Wearable Activity Tracker with Actigraphy for Sleep Evaluation and Circadian Rest-Activity Rhythm Measurement in Healthy Young Adults. Psychiatry Investig. 2017 Mar;14(2):179-185. doi: 10.4306/pi.2017.14.2.179. Epub 2017 Mar 6. PMID 28326116
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] http://www.thoracic.org/members/assemblies/assemblies/srn/questionaires/isi.php
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Gagnon C, Belanger L, Ivers H, Morin CM. Validation of the Insomnia Severity Index in primary care. J Am Board Fam Med. 2013 Nov-Dec;26(6):701-10. doi: 10.3122/jabfm.2013.06.130064. PMID 24204066
- [Background] http://www.nationalmssociety.org/For-Professionals/Researchers/Resources-for-Researchers/Clinical-Study-Measures/Multiple-Sclerosis-Quality-of-Life-Inventory-(MSQL
- [Background] Kurtzke JF. Rating neurologic impairment in multiple sclerosis: an expanded disability status scale (EDSS). Neurology. 1983 Nov;33(11):1444-52. doi: 10.1212/wnl.33.11.1444. PMID 6685237
- [Background] http://www.nationalmssociety.org/For-Professionals/Researchers/Resources-for-Researchers/Clinical-Study-Measures/Functional-Systems-Scores-(FSS)-and-Expanded-Disab
- [Background] https://scireproject.com/outcome-measures/outcome-measure-tool/ashworth-and-modified-ashworth-scale-mas/#1467983894080-2c29ca8d-88af
- [Background] http://www.thoracic.org/members/assemblies/assemblies/srn/questionaires/irls.php
- [Derived] Guarnaccia JB, Njike VY, Dutton A, Ayettey RG, Treu JA, Comerford BP, Sinha R. A pilot, randomized, placebo-controlled study of mindfulness meditation in treating insomnia in multiple sclerosis. BMC Neurol. 2023 Jul 11;23(1):263. doi: 10.1186/s12883-023-03309-0. PMID 37434109